CLINICAL TRIAL: NCT04232124
Title: Implementing the Los Angeles Barber - Pharmacist Model Hypertension Management in Nashville
Brief Title: Nashville - Hypertension Management Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of California, Los Angeles (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, David Harrison, Primary Investigator, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191470
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Execute a smaller version of the LA Barbershop BP Study through the new Nashville network as the test case for: A) recruiting regular patrons with uncontrolled HTN, B) conducting a research protocol and evaluating a HTN intervention; and C) creating a local registry of potential subjects as platform for enrolling black men in future research studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypertension Management Model (Experimental): Aim 1. Execute a smaller version of the LA Barbershop BP Study through the new Nashville network as the test case for: A) recruiting regular patrons with uncontrolled HTN, B) conducting a research protocol and evaluating a HTN intervention; and C) creating a local registry of potential subjects as platform for enrolling black men in future research studies.
  Interventions: Behavioral: Hypertension Management Model

INTERVENTIONS:
Behavioral: Hypertension Management Model — 1. Blood Pressure readings by barbers
  2. Clinical Pharmacist evaluation and counseling
  3. Blood pressure measurement
  4. Point of care basic metabolic panel measurement

SUMMARY:
Black men face a shorter life expectancy than white men due to poorer health outcomes associated with many chronic diseases, most notably hypertension and its cardiovascular complications. A lack of access to healthcare resources and poor engagement with healthcare providers drive these inequities. A seminal trial conducted in the Metro Los Angeles area demonstrated the effectiveness of using collaborative care partnerships between black-owned barbershops and pharmacists to reduce blood pressure in black men.

The purpose of this study is to test the feasibility and success of implementing a single-arm, smaller-scale version of the Los Angeles study in the Nashville area to provide additional empiric support for collaborative care partnerships to treat hypertension in other geographic locations.

DETAILED DESCRIPTION:
Uncontrolled hypertension (HTN) is a significant risk factor for mortality among non-Hispanic black men, and black men have the highest incidence of death from HTN of any race, ethnic, or gender group in the United States. Sustained, trusting interactions with healthcare professionals and a lack of access to healthcare resources are both significant drivers of these disparities. A cluster, randomized controlled trial in the Metro Los Angeles area demonstrated that health promotion by black barbers resulted in greater reductions in blood pressure (BP) when combined with medication management by specialty-trained pharmacists, as compared to health promotion by barbers alone.

The purposes of this single arm, pre-test/post-test study are to a) establish an effective network of barbershop research hubs in Nashville, b) test the feasibility of engaging with a specialty-trained pharmacist in collaboration with a barbershop to treat blood pressure in black men, and c) create a local registry of potential subjects as a platform for enrolling black men in future studies. There is no central hypothesis in this pilot implementation study, but the study will evaluate the ability of the barbershop-based research methodology to recruit and retain black men in a study; the fidelity to the intervention by barbers, the pharmacist, and the hypertensive male participants; and the effectiveness of the intervention on systolic blood pressure reduction and patient satisfaction. All participants will also be offered the opportunity to participate in a separate research registry for recruitment into future studies.

Research staff will offer free BP screening to all adult black men entering each shop for approximately 4 weeks, or until recruitment targets have been met. Patrons with a systolic BP > 140 mm Hg on two separate occasions will be eligible to participate. The patrons' existing physician or the lead physician or a study physician will sign a collaborative practice agreement for a specialty-trained pharmacist to provide care and prescribe BP medications within the study protocol. All participants in this study will execute a visit with the study physician for an evaluation to establish care, supported by the funding for this proposal.

Barbers will participate in training related to skills on BP measurement and counseling performed by either collaborating researchers from the University of California, Los Angeles-Cedars Sinai or from local study personnel. Barbers will frequently check and transmit the BP readings of their enrolled patrons and motivate them to work with the clinical pharmacist, who will meet them in their barbershops to optimize BP medication. The pharmacist will promote patient activation, intensify drug therapy under a collaborative practice agreement as permitted by Tennessee state law, send progress notes to the participant's physicians, and ensure appropriate safety monitoring after each medication change.

ELIGIBILITY:
Inclusion Criteria:

* Adults 35-79 years old
* Self - identify as Non-Hispanic black male
* Patron of one of the participating barbershops (4 haircuts in the last 6 months)
* Systolic BP> 140mm Hg on two screening days at least one day apart

Exclusion Criteria:

* Severe cognitive impairment
* Non-fluent in English
* Women
* Age < 35 years or > 79 years
* Systolic BP < 140 mm Hg at either screening
* Currently receiving chemotherapy for cancer
* Organ transplant patient
* Currently receiving dialysis
* Other conditions the physician investigator deem unsafe to participate
* Plans to move/relocate in next 12 months and/or travel out of area for > 1 month

Ages: 35 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study population is black men.
Enrollment: 30 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Harrison, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Vanderbilt University Medical Center, Nash, Tennessee
  - Masters Barbershop, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers with IRB approvals and also approved data sharing agreements contracts.
Supporting Information: Study Protocol, ICF
Time Frame: Data is currently available. It will remain available until the study is closed.
Access Criteria: IRB approval.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-Hispanic Black male clients, age 35-79 with systolic blood pressure > 140 mmHG on two screening visits. Enrolled participants were monitored closely throughout the 6-month study timeline and descriptive statistics preformed.
Groups:
- PharmD Community-based Delivery of Hypertension Management Including Medication Adjustment as Needed: Aim 1. Execute a smaller version of the LA Barbershop BP Study through the new Nashville network as the test case for: A) recruiting regular patrons with uncontrolled HTN, B) conducting a research protocol and evaluating a HTN intervention; and C) creating a local registry of potential subjects as platform for enrolling black men in future research studies.
  Hypertension Management Model: 1. Blood Pressure readings by barbers 2. Clinical Pharmacist evaluation and counseling 3. Blood pressure measurement 4. Point of care basic metabolic panel measurement
Period: Overall Study
Arm/Group | PharmD Community-based Delivery of Hypertension Management Including Medication Adjustment as Needed
Started | 30
Completed | 27
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Adults 35 - 79 years old, non-Hispanic black males, patron of one of the participating barbershops with Systolic BP > 140 on 2 screening visits.
Groups:
- Male Participants Who Received the Hypertension Management Model.: Adult Black males 39 to 79 years who were clients of one of our participating Barber Shops were screened for hypertension. Those with systolic BPs greater than 140 mmHg were asked to participate.
Arm/Group | Male Participants Who Received the Hypertension Management Model.
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Systolic Blood Pressure measurement, mmHg; Sitting position, average of three sequential measurements with an automated blood pressure monitor.
  mmHg | 157.7 (17.1)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Diastolic Blood Pressure measurement, mmHg; Sitting position, average of three sequential measurements with an automated blood pressure monitor.
  mmHg | 95.1 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic and Diastolic Blood Pressure
Description: Blood pressure changes were quantified as the baseline minus the 6 month value.
Time Frame: Baseline to 6 months
Population: Change in BP from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Male Participants Who Received the Hypertension Management Model
Number analyzed (Participants) | 27
mmHg
  Systolic | 21.1 (21.6)
  Diastolic | 19.5 (14.1)

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Description: Adverse events were assessed for participants once they signed their consent form. When a serious event was reported study personnel completed an adverse event form, submitted to the physician monitor for review and then submitted it to the DSMB if required.
Arm/Group | Male Participants Who Received the Hypertension Management Model
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Male Participants Who Received the Hypertension Management Model (N=30)
Seizure (Nervous system disorders) | 1 (1)
Transient Ischemic Attack (Blood and lymphatic system disorders) | 1 (1)
hyperglycemia (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Male Participants Who Received the Hypertension Management Model (N=30)
Covid Pneumonia (Immune system disorders) | 3 (3)
dizziness (Product Issues) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT04232124/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT04232124/ICF_000.pdf